CLINICAL TRIAL: NCT05880589
Title: Efficacy and Safety of Milk Secretory Supplement Containing Fenugreek, Banana Flower, and Ginger Extract in Breast-feeding Volunteers
Brief Title: Efficacy and Safety of Milk Secretory Supplement in Breast-feeding Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SIRB710/2565
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Lactation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Milk secretory supplement (Experimental): Milk secretory supplement composes of fenugreek, banana flower, ginger extract, docosahexaenoic acid, iron, folate, and iodine.
  Interventions: Dietary Supplement: Milk secretory supplement group
- Placebo group (Placebo Comparator): Placebo is tablet without fenugreek, banana flower, ginger extract, docosahexaenoic acid, iron, folate, and iodine.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Milk secretory supplement group — Take 2 tablet 2 times per day for 14 days
  Arms: Milk secretory supplement
Dietary Supplement: Placebo group — Take 2 tablet 2 times per day for 14 days
  Arms: Placebo group

SUMMARY:
The objective of this study are to evaluate efficacy and safety of milk secretory supplement containing fenugreek, banana flower, and ginger extract in breast-feeding volunteers

DETAILED DESCRIPTION:
There are 24 volunteers in this study. They are randomly divided into 2 groups which are milk secretory supplement group and placebo group. The volunteers take 2 tablets of the sample 2 times/day for 14 days. Amount of breast milk, calcium, iron, docosahexaenoic acid, quality of life, adverse reaction, and satisfaction before taking and after taking for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* During lactation
* Using only breast pump
* No taking medicine or dietary that has an effect on milk secretary including domperidone, banana flower, fenugreek, and ginger in 48 hours
* No smoking and alcohol drinking
* Can read and write in Thai language
* Can meet researcher at the date of appointment
* No complication after delivering

Exclusion Criteria:

* Have uncontrolled diseases, cancer, or heart disease
* Have immunocompromised disease or use steroid in 2 weeks
* Allergic to fenugreek, banana flower, ginger, docosahexaenoic acid, iron, folate, and iodine
* Cannot follow the protocol

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-11-10 (Estimated)

PRIMARY OUTCOMES:
Amount of breast milk | 14 days
  Measure volume of breast milk (ml) (High volume means high efficacy)

SECONDARY OUTCOMES:
Calcium in milk | 14 days
  Calcium in milk (mg/100ml) (High amount means high efficacy)
Iron in milk | 14 days
  Iron in milk (mg/100ml) (High amount means high efficacy)
Docosahexaenoic acid in milk | 14 days
  Docosahexaenoic acid in milk (g/100ml) (High amount means high efficacy)
Quality of life of volunteers | 14 days
  Use World Health Organization Quality of Life Brief - Thai questionnaire (0 to 4 scale means low to high quality of life)
Skin reaction after taking supplement | 14 days
  Found or not found
Gastrointestinal reaction after taking supplement | 14 days
  Found or not found
Respiratory tract reaction after taking supplement | 14 days
  Found or not found
Satisfaction after taking supplement | 14 days
  Use visual analogue scale (0 to 10 means lowest to highest satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Pornanong Aramwit, Professor, Principal Investigator — Chulalongkorn University
Locations (1):
- Pornanong Aramwit, Bangkok, Thailand